CLINICAL TRIAL: NCT01240577
Title: An Early Phase I Study of IPdR Absorption, Metabolism, and Safety in Patients With Advanced Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110026; 11-C-0026
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2013-02-26

CONDITIONS: Neoplasms; Lymphoma
Keywords: IPdR; Pharmacokinetics; Early Phase I; Cancer; Solid Tumor; Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — ropidoxuridine

INTERVENTIONS:
Drug: IPdR

SUMMARY:
Background:

- The experimental drug IPdR is broken down in the body to IdUrd, which has been given to patients to find out if it can improve radiation therapy. IdUrd has to be given through a vein; therefore this new drug (IPdR) has been made which can be taken by mouth. Researchers are interested in determining whether IPdR should also be studied to find out if it can improve radiation therapy. The current study is to find out if people absorb the drug given by mouth.

Objectives:

- To evaluate the levels of drug and its breakdown products in the blood following a single dose of IPdR by mouth. .

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with cancer (solid tumors or lymphomas) that have not responded to standard treatment.

Design:

* This study involves an initial dosing visit, one day of admission to the hospital for blood work, and a follow-up visit 14 days later.
* Participants will be screened with a physical examination and medical history, as well as blood and urine samples.
* Participants will receive a single dose of IPdR, and will provide multiple blood and urine samples for 24 hours after administration of the drug.
* Fourteen days after receiving IPdR, participants will have another physical examination and additional blood and urine tests to evaluate how IPdR has been broken down by the body.
* Cancer treatment will not be provided as part of this protocol.

DETAILED DESCRIPTION:
Background:

* The nucleoside analog iododeoxyuridine (IdUrd, NSC 39661) has shown promising activity as a radiosensitizer in preclinical models and has been evaluated in Phase I/II clinical trials. The extent of radiosensitization is directly related to the incorporation of IdUrd into tumor DNA as a replacement for thymidine.
* IPdR (NSC 726188) is an orally administered prodrug of IdUrd with a better therapeutic index in preclinical models.
* This first in human study of IPdR will evaluate whether IPdR is absorbed and what plasma levels of IPdR and its major metabolite, IdUrd, are achieved after a single oral dose.

Objectives:

* Measure plasma concentrations of IPdR, IdUrd, and IdUrd metabolites after a single oral dose of IPdR
* Determine the safety of administering a single oral dose of IPdR.

Eligibility:

-Patients must be greater than or equal to 18 years of age and have histologically confirmed solid tumors or lymphoid malignancies refractory to at least one line of standard treatment or for which no standard therapy is available. Patients should have adequate organ function and no disease-associated symptoms requiring immediate therapy or intervention.

Study Design:

* Patients will receive a single oral dose of IPdR on day 1.
* The initial IPdR dose will be 150 mg; dose escalation will be in 100% increments to a maximum of 2400 mg. One patient will be accrued to each dose level until we reach the highest dose level. Six patients will be accrued at dose level 5 (2400 mg).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically documented (confirmed at the Laboratory of Pathology, NCI) solid tumors or lymphoid malignancies that are refractory to at least one line of standard treatment or for which no standard therapy is available. Patients with lymphoid malignancies may be enrolled if they have disease for which standard therapy is currently not indicated. Patients should not have disease-associated symptoms requiring immediate therapy or intervention.
* Any prior chemotherapy or radiation therapy must have been completed greater than or equal to 2 weeks prior to enrollment (6 weeks for nitrosoureas or mitomycin C), and the patient must have recovered to eligibility levels from prior toxicity.
* Age greater than or equal to 18 years. Patients under 18 years of age are excluded because of their inability as a protected population to give appropriate consent to this non-therapeutic study.
* ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
* Life expectancy of at least 3 months.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/microL
  * platelets greater than or equal to 100,000/microL
  * total bilirubin less than 1.5 times institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) less than or equal to 3.0 times ULN
  * creatinine less than 1.5 times ULN

OR:

--creatinine clearance greater than or equal to 60 mL/min for patients with creatinine levels greater than or equal to 1.5 times ULN

* IPdR is a nucleoside analog and therefore potentially teratogenic. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 30 days after study drug administration. Because there is an unknown but potential risk for adverse events in nursing infants secondary to IPdR administration to the mother, nursing mothers should not receive IPdR.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, GI conditions limiting absorption, serious skin conditions, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or nursing.

INCLUSION OF WOMEN AND MINORITIES:

-Both men and women and members of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10-26; Primary Completion 2012-07-30 (Actual); Study Completion 2012-07-30 (Actual)

PRIMARY OUTCOMES:
-Measure plasma concentrations of IPdR, IdUrd, and IdUrd metabolites after a single oral dose of IPdR.-Determine the safety of administering a single oral dose of IPdR.

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schulz CA, Mehta MP, Badie B, McGinn CJ, Robins HI, Hayes L, Chappell R, Volkman J, Binger K, Arzoomanian R, Simon K, Alberti D, Feierabend C, Tutsch KD, Kunugi KA, Wilding G, Kinsella TJ. Continuous 28-day iododeoxyuridine infusion and hyperfractionated accelerated radiotherapy for malignant glioma: a phase I clinical study. Int J Radiat Oncol Biol Phys. 2004 Jul 15;59(4):1107-15. doi: 10.1016/j.ijrobp.2003.12.007. PMID 15234045
- [Background] Saif MW, Berk G, Cheng YC, Kinsella TJ. IPdR: a novel oral radiosensitizer. Expert Opin Investig Drugs. 2007 Sep;16(9):1415-24. doi: 10.1517/13543784.16.9.1415. PMID 17714027
- [Background] Kinsella TJ. An approach to the radiosensitization of human tumors. Cancer J Sci Am. 1996 Jul-Aug;2(4):184-93. PMID 9166528